CLINICAL TRIAL: NCT06764875
Title: A Randomized, Phase Ⅲ Study of Rilvegostomig in Combination With Fluoropyrimidine and Trastuzumab Deruxtecan Versus Trastuzumab, Chemotherapy, and Pembrolizumab for the First Line Treatment of HER2-positive Gastric Cancer (ARTEMIDE-Gastric01)
Brief Title: A Phase Ⅲ Study of Rilvegostomig in Combination With Fluoropyrimidine and Trastuzumab Deruxtecan as the First-line Treatment for HER2-positive Gastric Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D702AC00001; 2024-512583-57-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2024-12-12; First posted 2025-01-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: HER2-positive Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — trastuzumab deruxtecan; Trastuzumab; pembrolizumab; Fluorouracil; Capecitabine; Cisplatin; Oxaliplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will be conducted "Sponsor-blinded", such that intervention arm allocation is not known to Sponsor personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): T-DXd + Rilvegostomig + Fluoropyrimidine (Capecitabine OR 5-FU)
  Interventions: Drug: Rilvegostomig; Drug: Trastuzumab deruxtecan; Drug: 5-fluorouracil; Drug: Capecitabine
- Arm B (Active Comparator): Pembrolizumab + Trastuzumab + FP (5-FU plus cisplatin) or CAPOX (capecitabine plus oxaliplatin)
  Interventions: Drug: Trastuzumab; Drug: Pembrolizumab; Drug: 5-fluorouracil; Drug: Capecitabine; Drug: Cisplatin; Drug: Oxaliplatin
- Arm C (Active Comparator): Rilvegostomig + Trastuzumab + FP (5-FU plus cisplatin) or CAPOX (capecitabine plus oxaliplatin)
  Interventions: Drug: Rilvegostomig; Drug: Trastuzumab; Drug: 5-fluorouracil; Drug: Capecitabine; Drug: Cisplatin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Rilvegostomig — Q3W, intravenous infusion
  Other Names: AZD2936
  Arms: Arm A; Arm C
Drug: Trastuzumab deruxtecan — Q3W, intravenous infusion
  Other Names: T-DXd, DS-8201
  Arms: Arm A
Drug: Trastuzumab — Q3W, intravenous infusion
  Arms: Arm B; Arm C
Drug: Pembrolizumab — Q3W, intravenous infusion
  Arms: Arm B
Drug: 5-fluorouracil — Q3W, intravenous infusion
  Other Names: 5-FU
Drug: Capecitabine — BID, oral administration
Drug: Cisplatin — Q3W, intravenous infusion
  Arms: Arm B; Arm C
Drug: Oxaliplatin — Q3W, intravenous infusion
  Arms: Arm B; Arm C

SUMMARY:
This is a Phase Ⅲ, randomized, open-label, Sponsor-blinded, 3-arm, global, multicenter study assessing the efficacy and safety of rilvegostomig in combination with fluoropyrimidine and T-DXd (Arm A) compared to trastuzumab, chemotherapy, and pembrolizumab (Arm B) in HER2-positive locally advanced or metastatic gastric or GEJ adenocarcinoma participants whose tumors express PD L1 CPS ≥ 1. Rilvegostomig in combination with trastuzumab and chemotherapy will be evaluated in a separate arm (Arm C) to assess the contribution of each component in the experimental arm.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and safety of rilvegostomig in combination with fluoropyrimidine and T-DXd (Arm A) compared to trastuzumab, chemotherapy, and pembrolizumab (Arm B) in HER2-positive locally advanced or metastatic gastric or GEJ adenocarcinoma participants whose tumors express PD L1 CPS ≥ 1. Rilvegostomig in combination with trastuzumab and chemotherapy will be evaluated in a separate arm (Arm C) to assess the contribution of each component in the experimental arm.

This study will be conducted at up to 200-250 sites globally in approximately 25 countries.

ELIGIBILITY:
Inclusion Criteria:

* HER2 positive for gastric cancer on a tumor biopsy.
* PD-L1 combined positive score (CPS) ≥ 1.
* Provision of tumor tissue sample from recent biopsy adequate for HER2 and PD-L1 testing.
* Previously untreated, unresectable, locally advanced or metastatic gastric or GEJ adenocarcinoma.
* WHO or Eastern Cooperative Oncology Group performance status of 0 or 1.
* Have measurable target disease assessed by the Investigator based on RECIST v1.1.
* Have adequate organ and bone marrow function within 14 days before randomization.
* LVEF ≥ 55% within 28 days before randomization.
* Adequate treatment washout period before randomization.

Exclusion Criteria:

* Lack of physiological integrity of the upper gastrointestinal tract.
* Known dihydropyrimidine dehydrogenase enzyme deficiency.
* Contraindication to pembrolizumab or trastuzumab, contraindications to fluoropyrimidine (5-FU and capecitabine) or platinum (cisplatin and oxaliplatin) treatment as per local label.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease within 3 years before the first dose of study intervention and of low potential risk for recurrence.
* Persistent toxicities caused by previous anti-cancer therapy.
* Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring corticosteroid or anticonvulsant may be included in the study if they have recovered from the acute toxic effect of radiotherapy.
* Uncontrolled infection including tuberculosis and active hepatitis A infection.
* Uncontrolled infection requiring intravenous (IV) antibiotics, anti-virals, or antifungals.
* Recent receipt of live, attenuated vaccine.
* Chronic/active HBV or HCV infection unless controlled.
* Clinically significant cardiac or psychological conditions.
* Active or prior documented autoimmune or inflammatory disorders requiring chronic treatment with steroids or other immunosuppressive treatment.
* History of (non-infectious) ILD/pneumonitis, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Lung-specific intercurrent clinically significant illnesses.
* Any active non-infectious skin disease requiring systemic treatment.
* A pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or cell-free and concentrated ascites reinfusion therapy (CART).
* History of any of the following: drug-induced severe cutaneous adverse reaction.
* Any concurrent antic-ancer treatment with the exception of receptor activator of nuclear factor kappa-B ligand inhibitors.
* Have had major surgical procedure recently (excluding placement of vascular access) or recent significant traumatic injury or an anticipated need for major surgery during the study.
* Current or prior use of immunosuppressive medication within 14 days before study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2029-04-27 (Estimated); Study Completion 2030-12-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to approximately 6 years
  PFS is defined as time from randomization until progression per RECIST v1.1, or death due to any cause.
Overall Survival (OS) | Up to approximately 6 years
  OS is defined as time from randomization until the date of death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 6 years
  ORR according to RECIST v1.1. ORR is defined as the proportion of participants who have a complete response (CR) or partial response (PR).
Duration of Response (DoR) | Up to approximately 6 years
  DoR according to RECIST v1.1. DoR will be defined as the time from the date of first documented response until date of documented progression per RECIST v1.1 or death due to any cause.
Proportion of all randomized participants alive and progression-free at 6 months (PFS6) | Up to 6 months
  Proportion of all randomized participants alive and progression-free at 6 months calculated for progression.
Proportion of all randomized participants alive and progression-free at 12 months (PFS12) | Up to 12 months
  Proportion of all randomized participants alive and progression-free at 12 months calculated for progression.
Time to second progression or death (PFS2) | Up to approximately 6 years
  PFS2 is defined as the time from randomization to the earliest of the progression event (following the initial progression), after the first subsequent therapy, or death, where the first objective progression includes progression occurring after 2 missed visits.
Occurrence of adverse events (AEs) and serious adverse events (SAEs) | Up to approximately 6 years
  Occurrence of AEs and SAEs will be graded according to the revised NCI CTCAE v5.0.
Pharmacokinetics (PK) of rilvegostomig, T-DXd, total anti-HER2 antibody, DXd, 5-FU, and capecitabine in serum | Up to approximately 6 years
  Concentration of rilvegostomig, T-DXd, total anti-HER2 antibody, DXd, fluoropyrimidine, and capecitabine in serum or plasma.
Immunogenicity of rilvegostomig and T-DXd assessed by the presence of antidrug antibodies (ADAs) for rilvegostomig and T-DXd | Up to approximately 6 years
  Presence of antidrug antibodies (ADAs) for rilvegostomig and T-DXd (confirmatory results: titers and neutralizing antibodies for confirmed positive samples).
Increase in enteral feeding assistance and eating difficulties | Up to approximately 6 years
  Time to first-confirmed worsening of eating symptoms or initiation of feeding assistance among all participants, as randomized.
Proportion of time on study intervention with high side-effect bother | Up to approximately 6 years
  Proportion of time on study intervention with high side-effect bother relative to low side-effect burden as measured by the Patient Global Impression of Treatment Tolerability (PGI-TT).
Overall Survival at 12 months (OS12) | Up to 12 months
  Proportion of all randomized participants alive at 12 months.
Overall Survival at 24 months (OS24) | Up to 24 months
  Proportion of all randomized participants alive at 24 months.
Pharmacokinetics (PK) of rilvegostomig, T-DXd, total anti-HER2 antibody, DXd, 5-FU, and capecitabine in serum | Up to approximately 6 years
  PK parameters (peak and trough concentrations).

CONTACTS AND LOCATIONS:
Locations (238):
- United States (44):
  - Research Site, Anchorage, Alaska
  - Research Site, Phoenix, Arizona
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Santa Monica, California
  - Research Site, Solvang, California
  - Research Site, Upland, California
  - Research Site, Walnut Creek, California
  - Research Site, Aurora, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Niles, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Dyer, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Silver Spring, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Burnsville, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Reno, Nevada
  - Research Site, Summit, New Jersey
  - Research Site, Santa Fe, New Mexico
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Webster, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Charleston, West Virginia
  - Research Site, Madison, Wisconsin
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, Ciudad Autónoma Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Rosario
  - Research Site, Viedma
- Australia (4):
  - Research Site, Darlinghurst
  - Research Site, Heidelberg
  - Research Site, Murdoch
  - Research Site, Westmead
- Austria (4):
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wiener Neustadt
- Belgium (4):
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (9):
  - Research Site, Barretos
  - Research Site, Brasília
  - Research Site, Campo Grande
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Salvador
  - Research Site, São Paulo
  - Research Site, Vitória
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Barrie, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Montreal, Quebec
- Chile (5):
  - Research Site, Port Montt
  - Research Site, Rancagua
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (29):
  - Research Site, Anyang
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Linfen
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xining
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
- France (10):
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (14):
  - Research Site, Augsburg
  - Research Site, Bad Saarow
  - Research Site, Berlin
  - Research Site, Braunschweig
  - Research Site, Chemnitz
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Ludwigshafen
  - Research Site, Mannheim
  - Research Site, Ulm
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Gyöngyös
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Zalaegerszeg
- India (6):
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Varanasi
- Italy (8):
  - Research Site, Cagliari
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Rozzano
  - Research Site, Torino
  - Research Site, Tricase
- Japan (23):
  - Research Site, Akashi-shi
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Hiroshima
  - Research Site, Kasama-shi
  - Research Site, Kita-gun
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Matsuyama
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Ota-shi
  - Research Site, Sakaishi
  - Research Site, Sendai
  - Research Site, Shiwa-gun
  - Research Site, Suita-shi
  - Research Site, Sunto-gun
  - Research Site, Toyoake-shi
  - Research Site, Yokohama
- Malaysia (4):
  - Research Site, George Town
  - Research Site, Ipoh
  - Research Site, Kuala Lumpur
  - Research Site, Sabak Bernam
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Leiden
- Peru (4):
  - Research Site, Arequipa
  - Research Site, Callao
  - Research Site, Lima
  - Research Site, San Isidro
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Koszalin
  - Research Site, Olsztyn
  - Research Site, Przemyśl
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, Rio Piedras, Puerto Rico
- South Korea (5):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Gyeonggi-do
  - Research Site, Jeonnam
  - Research Site, Seoul
- Spain (7):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Ourense
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Banphaeo
  - Research Site, Dusit
  - Research Site, Khon Kaen
- Turkey (Türkiye) (7):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Diyarbakır
  - Research Site, Erzurum
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Mezitli
- United Kingdom (6):
  - Research Site, Cambridge
  - Research Site, Coventry
  - Research Site, Dundee
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Sutton
- Vietnam (5):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hồ Chí Minh
  - Research Site, Việt Trì
  - Research Site, Vinh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/